CLINICAL TRIAL: NCT00311948
Title: Telephone and Web-based Teen Tobacco Cessation in HMOs
Acronym: QWIThelper
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R01CA098685-02 (NIH); 1R01CA098685-01A2 (NIH)
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2006-09

CONDITIONS: Tobacco Use
Keywords: Teen smokers; Quithelper; Tobacco; Tobacco Website; Website Intervention; Tobacco counseling; Tobacco abstinence
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone counseling + interactive website (Active Comparator): Teen has access to interactive website and receives tailored telephone counseling
  Interventions: Behavioral: Telephone counseling + interactive website = more abstinence
- Control with interactive website (Other): Teen only has access to interactive website.
  Interventions: Behavioral: Behavioral: interactive website

INTERVENTIONS:
Behavioral: Telephone counseling + interactive website = more abstinence
  Arms: Telephone counseling + interactive website
Behavioral: Behavioral: interactive website
  Arms: Control with interactive website

SUMMARY:
The purpose of this study is to look at both the clinicians' ability to reach out to the teen smokers and to evaluate the efficacy of providing tobacco cessation support using a proactive telephone quitline combined with an interactive Web-based program for teens within a managed care environment.

DETAILED DESCRIPTION:
Health maintenance organizations have the mission, incentive, communication tools, and credibility with patients to reach out to teen members who use tobacco. The overall aim of this project is to refine and test both the potential reach and the efficacy of tobacco cessation support using a proactive telephone quitline combined with an interactive Web-based program for teens within a managed care environment. As part of a clinician-directed outreach effort, we will work closely with pediatric clinicians to maximize the program's reach into the teen smoker population as identified through the electronic data base of a large HMO. We will use letters and proactive outreach calls to assess current smoking status and recruit 600 15- to 18-year-old teen smokers who are interested in quitting and would be willing to receive cessation support via telephone and the Web. A second aim will be to randomly assign interested teen smokers to receive a proactive telephone- and Web-based tobacco cessation program or access to a website with cessation materials (control condition) to test the efficacy of the program on long-term cessation rates at 6- and 12-months. We will use several process measures to assess our ability to implement and consistently deliver both the telephone and Web components of the intervention. We will measure mediating variables to determine they support the hypothesized linkages between the theoretical constructs described by our cognitive behavioral model of action. An effective managed care partnership with clinicians to assess, recruit, and intervene with teen smokers would be of great interest to clinicians and health plan managers, highly exportable, and would be given high priority for implementation at the population level.

Our specific aims are as follows:

1. Compare the population-based recruitment yields and costs of three proactive outreach approaches: 1) outreach calls only to those teen smokers who are seen, advised, and referred to us by their clinician; 2) outreach calls to a random sample of teens shown as being smokers in the EMR; and 3) outreach calls to a sample of all teens
2. Assess efficacy/effectiveness in a randomized trial with 600 teen smokers to evaluate the hypothesis that proactive telephone-based counseling integrated with an interactive website will increase 6- and 12-month abstinence rates (30-day point prevalence) relative to a control condition receiving mailed cessation materials alone
3. Assess the hypothesis that the telephone and web-based intervention will improve longer-term maintenance of abstinence at an 12-month follow-up point compared to the control condition
4. Describe use patterns for key intervention process measures (e.g., calls completed, use of website) and determine if intervention affects outcome through theoretical mediators (e.g., pros/cons, stage, efficacy)
5. Determine the total costs of the telephone and web-based program from the perspective of the HMO and replication costs in other settings, and report costs as incremental costs per member per month, per program participant, and per quit.

ELIGIBILITY:
Inclusion Criteria:

* 15-18 years old
* both males and females
* smoking cigarettes at least four days a month
* some interest in quitting (will take all teen regardless of stage of readiness
* no evidence of treatment for depression, alcohol, or drugs in last year
* must consent
* have physician's approval for outreach to their panel
* have (or able to get) Internet access and phone access
* willingness to participate in study and follow-up procedures.

Exclusion Criteria:

* <15 years old
* >18 years old
* treated within 1 year for depression, alcohol, or drugs
* No internet access or phone access

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Actual)
Dates: Start 2006-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Participants' self-report of smoking one or more cigarettes in the past month at the 6-month and 12-month follow-up. | 6 months and 12 months
  self report of smoking in last 30 days
12-month measure to determine long-term assessment | 12-months
  Self report smoking or not smoking.

SECONDARY OUTCOMES:
A six-month assessment to determine short-term effects | 6 months
Assess the prevalence of smoking on 25 or more days per month | 1 month
Assess sustained abstinence (e.g., three and six months) at each follow-up, | 3 months and 6 months
  No smoking - yes or no at 3 month timeframe and 6 months timeframe
Assess change in stage of change | 6 months and 12 months
Assess amount smoked, and use of other tobacco products (including smokeless tobacco) in the last week, 30 days, three months, and six months prior to the follow-up assessment. | 30 days, 6 months, 12 months
Measure the proportion of teen smokers who are recruited through direct physician referral versus proactive outreach | 1 day
Compare the population-based recruitment yields and costs of three proactive outreach approaches that health plans might implement | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jack F Hollis, Ph.D., Principal Investigator — Kaiser Permanente
Locations (3):
- United States (3):
  - Oregon Research Institute, Eugene, Oregon
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Free & Clear, Inc., Seattle, Washington

REFERENCES:
- [Background] Committee on Substance Abuse. American Academy of Pediatrics: Tobacco's toll: implications for the pediatrician. Pediatrics. 2001 Apr;107(4):794-8. PMID 11335763
- [Background] Aveyard P, Cheng KK, Almond J, Sherratt E, Lancashire R, Lawrence T, Griffin C, Evans O. Cluster randomised controlled trial of expert system based on the transtheoretical ("stages of change") model for smoking prevention and cessation in schools. BMJ. 1999 Oct 9;319(7215):948-53. doi: 10.1136/bmj.319.7215.948. PMID 10514156
- [Background] Balch GI. Exploring perceptions of smoking cessation among high school smokers: input and feedback from focus groups. Prev Med. 1998 Sep-Oct;27(5 Pt 3):A55-63. doi: 10.1006/pmed.1998.0382. PMID 9808818
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Benuck I, Gidding SS, Binns HJ. Identification of adolescent tobacco users in a pediatric practice. Arch Pediatr Adolesc Med. 2001 Jan;155(1):32-5. doi: 10.1001/archpedi.155.1.32. PMID 11177059
- [Background] Bernard HR, Ryan GW. Text analysis: Qualitative and Quantitative Methods. In Handbook of Methods in Cultural Anthropology. Walnut Creek, CA: AltaMira Press; 1998
- [Background] Botvin GJ, Baker E, Dusenbury L, Tortu S, Botvin EM. Preventing adolescent drug abuse through a multimodal cognitive-behavioral approach: results of a 3-year study. J Consult Clin Psychol. 1990 Aug;58(4):437-46. doi: 10.1037//0022-006x.58.4.437. PMID 2212181
- [Background] Bowen DJ, Kinne S, Orlandi M. School policy in COMMIT: a promising strategy to reduce smoking by youth. J Sch Health. 1995 Apr;65(4):140-4. doi: 10.1111/j.1746-1561.1995.tb06217.x. PMID 7603051
- [Background] Bracken AC, Hersh AL, Johnson DJ. A computerized school-based health assessment with rapid feedback to improve adolescent health. Clin Pediatr (Phila). 1998 Nov;37(11):677-83. doi: 10.1177/000992289803701106. PMID 9825212
- [Background] Breslau N, Peterson EL. Smoking cessation in young adults: age at initiation of cigarette smoking and other suspected influences. Am J Public Health. 1996 Feb;86(2):214-20. doi: 10.2105/ajph.86.2.214. PMID 8633738
- [Background] Burt RD, Peterson AV Jr. Smoking cessation among high school seniors. Prev Med. 1998 May-Jun;27(3):319-27. doi: 10.1006/pmed.1998.0269. PMID 9612822
- [Background] Burton D. Tobacco cessation programs for adolescents. In: Richmond R, editor. Interventions for Smokers, an International Perspective. Baltimore, MD: Williams & Wilkins; 1994. p. 95-105.
- [Background] Cannell M. Generation Online: Internet use of teenagers. Science World 1999;55(9):5
- [Background] Chassin L, Presson CC, Rose JS, Sherman SJ. The natural history of cigarette smoking from adolescence to adulthood: demographic predictors of continuity and change. Health Psychol. 1996 Nov;15(6):478-84. doi: 10.1037//0278-6133.15.6.478. PMID 8973929
- [Background] Chen PH, White HR, Pandina RJ. Predictors of smoking cessation from adolescence into young adulthood. Addict Behav. 2001 Jul-Aug;26(4):517-29. doi: 10.1016/s0306-4603(00)00142-8. PMID 11456075
- [Background] Coambs RB, Li S, Kozlowski LT. Age interacts with heaviness of smoking in predicting success in cessation of smoking. Am J Epidemiol. 1992 Feb 1;135(3):240-6. doi: 10.1093/oxfordjournals.aje.a116277. PMID 1546699
- [Background] Curry SJ, Grothaus LC, McAfee T, Pabiniak C. Use and cost effectiveness of smoking-cessation services under four insurance plans in a health maintenance organization. N Engl J Med. 1998 Sep 3;339(10):673-9. doi: 10.1056/NEJM199809033391006. PMID 9725926
- [Background] Curry SJ, McBride C, Grothaus LC, Louie D, Wagner EH. A randomized trial of self-help materials, personalized feedback, and telephone counseling with nonvolunteer smokers. J Consult Clin Psychol. 1995 Dec;63(6):1005-14. doi: 10.1037//0022-006x.63.6.1005. PMID 8543703
- [Background] Dent CW, Sussman S, Stacy AW, Craig S, Burton D, Flay BR. Two-year behavior outcomes of project towards no tobacco use. J Consult Clin Psychol. 1995 Aug;63(4):676-7. doi: 10.1037//0022-006x.63.4.676. PMID 7673547
- [Background] Department of Commerce. Falling Through the Net: Defining the Digital Divide, 1999; Online at http://www.ntia.doc.gov/ntiahome/fttn99/contents.html. Last viewed January, 2002.
- [Background] Digiusto E. Pros and cons of cessation interventions for adolescent smokers at school. In R Richmond (ed). Interventions for smokers: An international perspective. Baltimore: MD: Williams & Wilkins;107 136, 1994.
- [Background] Drummond MF, O'Brien B, Stoddart GL, Torrance GW. Methods for the Economic Evaluation of Health Care Programmes. 2nd Edition. Oxford: Oxford University Press, 1997.
- [Background] Elder JP, Wildey M, de Moor C, Sallis JF Jr, Eckhardt L, Edwards C, Erickson A, Golbeck A, Hovell M, Johnston D, et al. The long-term prevention of tobacco use among junior high school students: classroom and telephone interventions. Am J Public Health. 1993 Sep;83(9):1239-44. doi: 10.2105/ajph.83.9.1239. PMID 8362998
- [Background] Engels RC, Knibbe RA, de Vries H, Drop MJ. Antecedents of smoking cessation among adolescents: who is motivated to change? Prev Med. 1998 May-Jun;27(3):348-57. doi: 10.1006/pmed.1998.0304. PMID 9612825
- [Background] A clinical practice guideline for treating tobacco use and dependence: A US Public Health Service report. The Tobacco Use and Dependence Clinical Practice Guideline Panel, Staff, and Consortium Representatives. JAMA. 2000 Jun 28;283(24):3244-54. PMID 10866874
- [Background] Flay BR, Hu FB, Richardson J. Psychosocial predictors of different stages of cigarette smoking among high school students. Prev Med. 1998 Sep-Oct;27(5 Pt 3):A9-18. doi: 10.1006/pmed.1998.0380. PMID 9808813
- [Background] Fleiss JL. Statistical methods for rates and proportions. Second Ed. New York: John Wiley & Sons; 1981.
- [Background] Flynn BS, Worden JK, Secker-Walker RH, Pirie PL, Badger GJ, Carpenter JH. Long-term responses of higher and lower risk youths to smoking prevention interventions. Prev Med. 1997 May-Jun;26(3):389-94. doi: 10.1006/pmed.1997.0159. PMID 9144764
- [Background] Glasgow RE, Mullooly JP, Vogt TM, Stevens VJ, Lichtenstein E, Hollis JF, Lando HA, Severson HH, Pearson KA, Vogt MR. Biochemical validation of smoking status: pros, cons, and data from four low-intensity intervention trials. Addict Behav. 1993 Sep-Oct;18(5):511-27. doi: 10.1016/0306-4603(93)90068-k. PMID 8310871
- [Background] Glasgow RE, Toobert DJ, Hampson SE. Effects of a brief office-based intervention to facilitate diabetes dietary self-management. Diabetes Care. 1996 Aug;19(8):835-42. doi: 10.2337/diacare.19.8.835. PMID 8842601
- [Background] Glasgow RE, La Chance PA, Toobert DJ, Brown J, Hampson SE, Riddle MC. Long-term effects and costs of brief behavioural dietary intervention for patients with diabetes delivered from the medical office. Patient Educ Couns. 1997 Nov;32(3):175-84. doi: 10.1016/s0738-3991(97)00039-6. PMID 9423499
- [Background] Glasgow RE, Fisher EB, Anderson BJ, LaGreca A, Marrero D, Johnson SB, Rubin RR, Cox DJ. Behavioral science in diabetes. Contributions and opportunities. Diabetes Care. 1999 May;22(5):832-43. doi: 10.2337/diacare.22.5.832. PMID 10332691
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Glasgow RE, Wagner EH, Kaplan RM, Vinicor F, Smith L, Norman J. If diabetes is a public health problem, why not treat it as one? A population-based approach to chronic illness. Ann Behav Med. 1999 Spring;21(2):159-70. doi: 10.1007/BF02908297. PMID 10499137
- [Background] Glasgow RE, Eakin EG. Medical office-based interventions. In: Snoek FJ, Skinner CS., Eds. Psychological Aspects of Diabetes Care. New York: John Wiley and Sons; 2000
- [Background] Gold MR, Siegel JE, Russell LB, Weinstein MC. Cost-Effectiveness in Health and Medicine. New York: Oxford University Press, 1996.
- [Background] Richard L, Breton ER, Lehoux P, Martin C, Roy D. [Public health professionals' perceptions regarding two dimensions of health promotion: the ecological approach and community participation]. Can J Public Health. 1999 Mar-Apr;90(2):99-103. doi: 10.1007/BF03404110. French. PMID 10349215
- [Background] Grzywacz JG, Fuqua J. The social ecology of health: leverage points and linkages. Behav Med. 2000 Fall;26(3):101-15. doi: 10.1080/08964280009595758. PMID 11209591
- [Background] Hines D. Young smokers' attitudes about methods for quitting smoking: barriers and benefits to using assisted methods. Addict Behav. 1996 Jul-Aug;21(4):531-5. doi: 10.1016/0306-4603(95)00076-3. PMID 8830912
- [Background] Hollis JF, Bills R, Whitlock E, Stevens VJ, Mullooly J, Lichtenstein E. Implementing tobacco interventions in the real world of managed care. Tob Control. 2000;9 Suppl 1(Suppl 1):I18-24. doi: 10.1136/tc.9.suppl_1.i18. No abstract available. PMID 10688926
- [Background] Hollis JF, Lichtenstein E, Mount K, Vogt TM, Stevens VJ. Nurse-assisted smoking counseling in medical settings: minimizing demands on physicians. Prev Med. 1991 Jul;20(4):497-507. doi: 10.1016/0091-7435(91)90047-8. PMID 1871078
- [Background] Hollis JF, Lichtenstein E, Vogt TM, Stevens VJ, Biglan A. Nurse-assisted counseling for smokers in primary care. Ann Intern Med. 1993 Apr 1;118(7):521-5. doi: 10.7326/0003-4819-118-7-199304010-00006. PMID 8442622
- [Background] Hollis JF, Polen MR, Lichtenstein E, Whitlock EP. Tobacco use patterns and attitudes among teens being seen for routine primary care. Am J Health Promot. 2003 Mar-Apr;17(4):231-9. doi: 10.4278/0890-1171-17.4.231. PMID 12640779
- [Background] Hollis JF, Vogt TM, Stevens VJ, Biglan A, Severson H, Lichtenstein E. The Tobacco Reduction and Cancer Control (TRACC) Program: Team approaches to counseling in medical and dental settings. In US Department of Health and Human Services, Tobacco and the Clinician: Interventions for Medical and Dental Practice, pp. 143 185. Smoking and Tobacco Control: Monograph 5. US Department of Health and Human Services, Public Health Service, National Institutes of Health. NIH Publication No. 94 3693, January 1994.
- [Background] Hu TW, Lin Z, Keeler TE. Teenage smoking, attempts to quit, and school performance. Am J Public Health. 1998 Jun;88(6):940-3. doi: 10.2105/ajph.88.6.940. PMID 9618625
- [Background] Jaen CR, Stange KC, Tumiel LM, Nutting P. Missed opportunities for prevention: smoking cessation counseling and the competing demands of practice. J Fam Pract. 1997 Oct;45(4):348-54. PMID 9343057
- [Background] Klein JD. Incorporating effective smoking prevention and cessation counseling into practice. Pediatr Ann. 1995 Dec;24(12):646-52. doi: 10.3928/0090-4481-19951201-08. No abstract available. PMID 8747707
- [Background] Klein JD, Levine LJ, Allan MJ. Delivery of smoking prevention and cessation services to adolescents. Arch Pediatr Adolesc Med. 2001 May;155(5):597-602. doi: 10.1001/archpedi.155.5.597. PMID 11343505
- [Background] Kottke TE, Battista RN, DeFriese GH, Brekke ML. Attributes of successful smoking cessation interventions in medical practice. A meta-analysis of 39 controlled trials. JAMA. 1988 May 20;259(19):2883-9. doi: 10.1001/jama.259.19.2883. PMID 3367456
- [Background] Lamb JM, Albrecht SA, Sereika S. Consideration of factors prior to implementing a smoking cessation program. J Sch Nurs. 1998 Feb;14(1):14-9. PMID 9505644
- [Background] Lamkin LP, Houston TP. Nicotine dependency and adolescents: preventing and treating. Prim Care. 1998 Mar;25(1):123-35. doi: 10.1016/s0095-4543(05)70328-6. PMID 9469919
- [Background] Lichtenstein E, Glasgow RE, Lando HA, Ossip-Klein DJ, Boles SM. Telephone counseling for smoking cessation: rationales and meta-analytic review of evidence. Health Educ Res. 1996 Jun;11(2):243-57. doi: 10.1093/her/11.2.243. PMID 10163409
- [Background] Institute of Medicine (US) Committee on Preventing Nicotine Addiction in Children and Youths; Lynch BS, Bonnie RJ, editors. Growing up Tobacco Free: Preventing Nicotine Addiction in Children and Youths. Washington (DC): National Academies Press (US); 1994. Available from http://www.ncbi.nlm.nih.gov/books/NBK236763/ PMID 25144107
- [Background] McAfee T, Wilson J, Dacey S, Sofian N, Curry S, Wagener B. Awakening the sleeping giant: mainstreaming efforts to decrease tobacco use in an HMO. HMO Pract. 1995 Sep;9(3):138-43. PMID 10151099
- [Background] McIlvain HE, Crabtree BF, Gilbert C, Havranek R, Backer EL. Current trends in tobacco prevention and cessation in Nebraska physicians' offices. J Fam Pract. 1997 Feb;44(2):193-202. PMID 9040523
- [Background] Miller WL, Crabtree BF. Clinical research. In: Handbook of Qualitative Research. NK Denzin & YS Lincoln (eds.) Thousand Oaks, CA: Sage Publications; 1994.
- [Background] Miller WR, Rollnick S. Motivational Interviewing: Preparing People to Change Addictive Behavior. New York: The Guilford Press; 1991.
- [Background] Moolchan ET, Ernst M, Henningfield JE. A review of tobacco smoking in adolescents: treatment implications. J Am Acad Child Adolesc Psychiatry. 2000 Jun;39(6):682-93. doi: 10.1097/00004583-200006000-00006. PMID 10846302
- [Background] Morgan DL, ed. The Focus Group Guidebook. Thousand Oaks, CA: Sage; 1998.
- [Background] National Cancer Institute. Scientific priorities for cancer research: NCI's extraordinary opportunities. Online at: http://2001.cancer.gov/communications.htm. Last viewed: January 2002.
- [Background] Nielsen NetRatings. (2001, May) [On-line]. http://www.eratings.com/news/20010430.htm. Report available at: http://www.nwcn.com/cybernews/329373_TSportlandwired040301.html
- [Background] Nichter M, Nichter M, Vuckovic N, Quintero G, Ritenbaugh C. Smoking experimentation and initiation among adolescent girls: qualitative and quantitative findings. Tob Control. 1997 Winter;6(4):285-95. doi: 10.1136/tc.6.4.285. PMID 9583626
- [Background] Nichter M, Vuckovic N, Parker S. The looking good, feeling good program: A multi-ethnic intervention for healthy body image, nutrition and physical activity. In Preventing Eating Disorders: A Handbook of Intervention and Special Challenges. E Piran, MP Levine and C Steiner-Adair, eds. Philadelphia: Brunner-Mozel; 1999, 173-93.
- [Background] O'Connor EA, Hollis JF, Polen MR, Lichtenstein E. Adolescent health care visits: opportunities for brief prevention messages. Eff Clin Pract. 1999 Nov-Dec;2(6):272-6. PMID 10788025
- [Background] Oregon Youth Risk Behavior Survey. Health Division, Oregon Department of Human Resources. Portland, Oregon, Dec. 1993.
- [Background] Orleans CT, Schoenbach VJ, Wagner EH, Quade D, Salmon MA, Pearson DC, Fiedler J, Porter CQ, Kaplan BH. Self-help quit smoking interventions: effects of self-help materials, social support instructions, and telephone counseling. J Consult Clin Psychol. 1991 Jun;59(3):439-48. doi: 10.1037//0022-006x.59.3.439. PMID 2071729
- [Background] Paavola M, Vartiainen E, Puska P. Smoking cessation between teenage years and adulthood. Health Educ Res. 2001 Feb;16(1):49-57. doi: 10.1093/her/16.1.49. PMID 11252283
- [Background] Pallonen UE, Velicer WF, Prochaska JO, Rossi JS, Bellis JM, Tsoh JY, Migneault JP, Smith NF, Prokhorov AV. Computer-based smoking cessation interventions in adolescents: description, feasibility, and six-month follow-up findings. Subst Use Misuse. 1998 Mar;33(4):935-65. doi: 10.3109/10826089809056250. PMID 9548631
- [Background] Pallonen UE, Prochaska JO, Velicer WF, Prokhorov AV, Smith NF. Stages of acquisition and cessation for adolescent smoking: an empirical integration. Addict Behav. 1998 May-Jun;23(3):303-24. doi: 10.1016/s0306-4603(97)00074-9. PMID 9668929
- [Background] Perry CL, Griffin G, Murray DM. Assessing needs for youth health promotion. Prev Med. 1985 May;14(3):379-93. doi: 10.1016/0091-7435(85)90064-7. PMID 4059190
- [Background] Peterson AV Jr, Kealey KA, Mann SL, Marek PM, Sarason IG. Hutchinson Smoking Prevention Project: long-term randomized trial in school-based tobacco use prevention--results on smoking. J Natl Cancer Inst. 2000 Dec 20;92(24):1979-91. doi: 10.1093/jnci/92.24.1979. PMID 11121460
- [Background] Pew Internet & American Life Project. The Internet and Education: Findings of the Pew Internet & American Life Project. Online at: http://www.pewinternet.org/reports/toc.asp?Report=39. Last viewed: January 2002
- [Background] Plummer BA, Velicer WF, Redding CA, Prochaska JO, Rossi JS, Pallonen UE, Meier KS. Stage of change, decisional balance, and temptations for smoking: measurement and validation in a large, school-based population of adolescents. Addict Behav. 2001 Jul-Aug;26(4):551-71. doi: 10.1016/s0306-4603(00)00144-1. PMID 11456077
- [Background] Prince F. The relative effectiveness of a peer-led and adult-led smoking intervention program. Adolescence. 1995 Spring;30(117):187-94. PMID 7625255
- [Background] Prochaska JO, DiClemente CC, Norcross JC. In search of how people change. Applications to addictive behaviors. Am Psychol. 1992 Sep;47(9):1102-14. doi: 10.1037//0003-066x.47.9.1102. PMID 1329589
- [Background] Prochaska JO, DiClemente CC, Velicer WF, Ginpil S, Norcross JC. Predicting change in smoking status for self-changers. Addict Behav. 1985;10(4):395-406. doi: 10.1016/0306-4603(85)90036-x. PMID 4091072
- [Background] Prochaska JO, DiClemente CC. Stages and processes of self-change of smoking: toward an integrative model of change. J Consult Clin Psychol. 1983 Jun;51(3):390-5. doi: 10.1037//0022-006x.51.3.390. No abstract available. PMID 6863699
- [Background] Roberts DF, Foehr UB, Rideout VJ, Brodie M. Kids, Media @ The New Millennium. A Kaiser Family Foundation Report, November; 1999.
- [Background] Rost K, Burnam MA, Smith GR. Development of screeners for depressive disorders and substance disorder history. Med Care. 1993 Mar;31(3):189-200. doi: 10.1097/00005650-199303000-00001. PMID 8450677
- [Background] Sargent JD, Mott LA, Stevens M. Predictors of smoking cessation in adolescents. Arch Pediatr Adolesc Med. 1998 Apr;152(4):388-93. doi: 10.1001/archpedi.152.4.388. PMID 9559717
- [Background] Secker-Walker RH, Worden JK, Holland RR, Flynn BS, Detsky AS. A mass media programme to prevent smoking among adolescents: costs and cost effectiveness. Tob Control. 1997 Autumn;6(3):207-12. doi: 10.1136/tc.6.3.207. PMID 9396105
- [Background] Senn S. Testing for baseline balance in clinical trials. Stat Med. 1994 Sep 15;13(17):1715-26. doi: 10.1002/sim.4780131703. PMID 7997705
- [Background] Siqueira LM, Rolnitzky LM, Rickert VI. Smoking cessation in adolescents: the role of nicotine dependence, stress, and coping methods. Arch Pediatr Adolesc Med. 2001 Apr;155(4):489-95. doi: 10.1001/archpedi.155.4.489. PMID 11296077
- [Background] Smith TA, House RF Jr, Croghan IT, Gauvin TR, Colligan RC, Offord KP, Gomez-Dahl LC, Hurt RD. Nicotine patch therapy in adolescent smokers. Pediatrics. 1996 Oct;98(4 Pt 1):659-67. PMID 8885942
- [Background] SRNT Subcommittee on Biochemical Verification. Biochemical verification of tobacco use and cessation. Nicotine Tob Res. 2002 May;4(2):149-59. doi: 10.1080/14622200210123581. No abstract available. PMID 12028847
- [Background] Solas V.3.0. Cork, Ireland; Statistical Solutions Ltd., 2001.
- [Background] Strecher VJ. Computer-tailored smoking cessation materials: a review and discussion. Patient Educ Couns. 1999 Feb;36(2):107-17. doi: 10.1016/s0738-3991(98)00128-1. PMID 10223016
- [Background] Sussman S. Effects of sixty six adolescent tobacco use cessation trials and seventeen prospective studies of self-initiated quitting. Tob Induc Dis. 2002 Jan 15;1(1):35-81. doi: 10.1186/1617-9625-1-1-35. PMID 19570247
- [Background] Sussman S, Dent CW, Stacy AW, Sun P, Craig S, Simon TR, Burton D, Flay BR. Project towards no tobacco use: 1-year behavior outcomes. Am J Public Health. 1993 Sep;83(9):1245-50. doi: 10.2105/ajph.83.9.1245. PMID 8362999
- [Background] Sussman S, Lichtman K, Ritt A, Pallonen UE. Effects of thirty-four adolescent tobacco use cessation and prevention trials on regular users of tobacco products. Subst Use Misuse. 1999 Sep;34(11):1469-503. doi: 10.3109/10826089909039411. PMID 10468104
- [Background] Sussman S, Dent CW, Severson H, Burton D, Flay BR. Self-initiated quitting among adolescent smokers. Prev Med. 1998 Sep-Oct;27(5 Pt 3):A19-28. doi: 10.1006/pmed.1998.0379. PMID 9808814
- [Background] The Kaiser Family Foundation. Generation Rx.com How Young people Use the Internet for Health Information. Online at: http://www.kff.org/content/2001/20011211a/. 2001. Last viewed January 2002.
- [Background] Thorndike AN, Ferris TG, Stafford RS, Rigotti NA. Rates of U.S. physicians counseling adolescents about smoking. J Natl Cancer Inst. 1999 Nov 3;91(21):1857-62. doi: 10.1093/jnci/91.21.1857. PMID 10547392
- [Background] US Department of Health and Human Services. Preventing Tobacco Use Among Young People: A Report of the Surgeon General. Atlanta, Georgia: US Department of Health and Human Services, Public Health Service, Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion, Office on Smoking and Health; 1994.
- [Background] Velicer WF, Prochaska JO, Rossi JS, Snow MG. Assessing outcome in smoking cessation studies. Psychol Bull. 1992 Jan;111(1):23-41. doi: 10.1037/0033-2909.111.1.23. PMID 1539088
- [Background] Vuckovic N, Polen MR, Hollis JF. The problem is getting us to stop. What teens say about smoking cessation. Prev Med. 2003 Sep;37(3):209-18. doi: 10.1016/s0091-7435(03)00115-4. PMID 12914826
- [Background] Woodruff SI, Edwards CC, Conway TL, Elliott SP. Pilot test of an Internet virtual world chat room for rural teen smokers. J Adolesc Health. 2001 Oct;29(4):239-43. doi: 10.1016/s1054-139x(01)00262-2. PMID 11587907
- [Background] Worden JK, Flynn BS, Solomon LJ, Secker-Walker RH, Badger GJ, Carpenter JH. Using mass media to prevent cigarette smoking among adolescent girls. Health Educ Q. 1996 Nov;23(4):453-68. doi: 10.1177/109019819602300406. PMID 8910024
- [Background] Zapka JG, Fletcher K, Pbert L, Druker SK, Ockene JK, Chen L. The perceptions and practices of pediatricians: tobacco intervention. Pediatrics. 1999 May;103(5):e65. doi: 10.1542/peds.103.5.e65. PMID 10224209
- [Background] Zhu SH, Sun J, Billings SC, Choi WS, Malarcher A. Predictors of smoking cessation in U.S. adolescents. Am J Prev Med. 1999 Apr;16(3):202-7. doi: 10.1016/s0749-3797(98)00157-3. PMID 10198659